CLINICAL TRIAL: NCT05027334
Title: A Mobile System Framework to Support the Autonomous Self-management of Pre-diabetes and Type 2 Diabetes Mellitus Patients in Mauritius
Brief Title: Self-Management of Type-2 Diabetes Using a Mobile Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mauritius (Other)
Responsible Party: Principal Investigator, Abha Jodheea-Jutton, Dr, University of Mauritius
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UoM/R213
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus, E health, glycaemic control, physical activity
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Participants will be asked to use a designed mobile app to monitor their blood sugar levels
  Interventions: Other: DiaMon - Mobile Application for Type 2 Diabetes mellitus and pre-diabetes

INTERVENTIONS:
Other: DiaMon - Mobile Application for Type 2 Diabetes mellitus and pre-diabetes — Each participant will be provided with a mobile application aimed at monitoring their clinical markers such as FBG and HbA1c. The mobile application consists of medical details and demographics as well as a section dedicated to daily glucose levels and record of physical activity.

SUMMARY:
Diabetes Mellitus (DM) is a global health emergency, since its prevalence has become alarming in many countries in the previous years. Because of the increasing healthcare requirement, it has also progressively become an economic burden for every country. From the International Diabetes Federation (IDF) Atlas (International Diabetes Federation, 2015), 415 million people worldwide were estimated to have DM in 2015 and this figure is expected to rise to 642 million in 2040. DM contributed to 5 million adult deaths globally in 2015. Mauritius has one of the highest DM prevalence in the world (24.3% prevalence for ages 20 - 79) for 2015 (International Diabetes Federation, 2015). 2,932 adult died due to Diabetes, and the average cost of DM related problems amount to 2 billion rupees per year. The Mauritius Non Communicable Diseases Survey (Ministry of Health and Quality of Life, 2015) reports an estimated 257,442 people between the ages of 25 and 74 with Diabetes in Mauritius. A high prevalence of pre-diabetes is also noted, which may subsequently result in diabetes and heart disease, if not appropriately managed. The DM epidemic has a significant impact locally and globally, calling for urgent remedial strategies to curb the spread.

Studies have shown that patient's self-care including monitoring of blood glucose improve glycemic control (Allemann et al, 2009; Skeie et al, 2009; Istepanian et al, 2009). Patients are currently empowered through face to face counselling, websites, social media and other state of the art technologies. The use of smart phones for self-monitoring of blood glucose has shown to have substantial beneficial effects (Liang et al, 2011; Pal et al 2014). This project aims at using mobile technologies to instil behavioural changes in people living with DM and pre-diabetes in an attempt to alleviate the long term problems associated with DM. More precisely, it will constitute the development of an autonomous system for self-management of type 2 diabetes mellitus (T2DM) patients in Mauritius. The prototype will be tested for feasibility among patients with T2DM and pre-diabetes. It is expected that the proposed system will help to reduce the financial burden on the healthcare system in Mauritius through patient empowerment and improved self-care in the long run.

DETAILED DESCRIPTION:
he global burden of diabetes mellitus is an issue of increasing concern globally. The social and economic burden is soaring, pushing scientist to discover alternative options to reduce the burden. It is estimated that the burden is worse in countries with limited resources such as Mauritius.

Mauritius has one of the highest DM prevalence in the world (24.3% prevalence for ages 20 - 79) for 2015 (International Diabetes Federation, 2015). 2,932 adult died due to diabetes, and the average cost of DM related problems amount to 2 billion rupees per year. The Mauritius Non Communicable Diseases Survey (Ministry of Health and Quality of Life, 2015) reports an estimated 257,442 people between the ages of 25 and 74 with Diabetes in Mauritius. A high prevalence of pre-diabetes is also noted, which may subsequently result in diabetes and heart disease, if not appropriately managed. The DM epidemic has a significant impact locally and globally, calling for urgent remedial strategies to curb the spread.

Studies have shown that patient's self-care including monitoring of blood glucose improve glycemic control (Allemann et al, 2009; Skeie et al, 2009; Istepanian et al, 2009). Patients are currently empowered through face to face counselling, websites, social media and other state of the art technologies. The use of smart phones for self-monitoring of blood glucose has shown to have substantial beneficial effects (Liang et al, 2011; Pal et al 2014).

Aims and objectives:

The aim of the study is to evaluate the effect on glycaemic levels among patients living with type 2 diabetes who are using a newly designed mobile application.

The objectives are to:

Measure the change in HbA1c after 3 months of using the application Compare secondary outcomes such as weight and BMI following the use of the application Assess the perception of patients using the digital tool and relate behavioural changes with the use of the application

Methodology:

A single arm prospective non randomised study is proposed. Participants will be recruited using adverts in the local newspapers and social media. Interested participants will be screened for eligibility and given the mobile application to use. They will be advised to record their daily fasting and post-prandial blood glucose as well as their levels of physical activity.

The following clinical and biomarkers will be checked before and after the use of the intervention: HbA1c, FBS, weight, BMI and blood pressure. The duration of follow up will be 3-6 months. An investigator designed questionnaire will be used to evaluate the use of the mobile app.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HbA1c 7-8% (stable T2DM) Patients with Impaired fasting glucose or impaired glucose tolerance Patients between 18 -74 years Both males and female patients Participants diagnosed with T2DM Participants able to provide consent Participants able to use the SMART phones

Exclusion Criteria:

* Patients with HbA1c >9% (poorly controlled DM) Patients with type 1 diabetes mellitus Pregnant women Patients with gestational DM Patients unable to use smart devices Patients unable to provide consent People with other chronic diseases or health problems which can interfere with glycaemic control (e.g brittle asthma/COPD and using oral steroids)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Glycaemic control | 3 months
  The glycaemic control was measured through glycated haemoglobin (HbA1c)
Fasting blood glucose (FBG) | 3 months
  FBG was measured on a daily basis and a reduction in FBG was sought.

SECONDARY OUTCOMES:
Weight | 3 months
  a change in weight was measured through measurement of weight before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Abha Jodheea-Jutton, Principal Investigator — University of Mauritius
Locations (1):
- University of Mauritius, Réduit, Moka District, Mauritius

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant Data has been recorded in an anonymous format digitally and is available upon request.